CLINICAL TRIAL: NCT02823405
Title: A Phase 1b Trial of X4P-001 Alone and With Pembrolizumab in Patients With Advanced Melanoma
Brief Title: X4P-001 and Pembrolizumab in Patients With Advanced Melanoma
Acronym: X4P-001-MELA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-MELA
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Melanoma
Keywords: Advance malignancy
MeSH Terms: conditions — Melanoma | interventions — mavorixafor; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- X4P-001 + Pembrolizumab (Experimental): X4P-001 alone, then adding pembrolizumab
  Interventions: Drug: X4P-001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: X4P-001 — X4P-001 100 mg capsules, administered orally, continuous daily dosing
  Other Names: AMD11070
Drug: Pembrolizumab — Pembrolizumab 2 mg/kg, administered by IV infusion every 3 weeks
  Other Names: Keytruda

SUMMARY:
The goals of this protocol are 1) to investigate the safety and tolerability of X4P-001 in combination with Keytruda® (pembrolizumab) in patients with advanced melanoma, and 2) to assess serial biopsies of melanoma tumor lesions obtained throughout the study for inflammatory and tumor cell infiltrates. After completion of study treatment, participants with resectable disease will undergo surgery, unresectable participants may continue on pembrolizumab as standard of care.

DETAILED DESCRIPTION:
X4P-001 is an orally bioavailable CXCR4 antagonist that has demonstrated activity in various tumor models. CXCR4 (C-X-C chemokine receptor type 4) is the receptor for CXCL12 (C-X-C chemokine ligand type 12). CXCL12 has potent chemotactic activity for lymphocytes and MDSCs (myeloid-derived suppressor cells), and is important in homing of hematopoietic stem cells to the bone marrow. CXCR4 is also expressed and active on multiple types of human cancers, including melanoma, ccRCC, and ovarian cancer. Additionally, increased expression of CXCR4 on tumor cells has been associated with significantly decreased overall participant survival.

In animal cancer models, interference with CXCR4 function has been demonstrated to disrupt the tumor microenvironment (TME) and unmask the tumor to immune attack by multiple mechanisms, including:

* Decreasing the infiltration of MDSCs
* Increasing the ratio of CD8+ T cells to Treg cells
* Eliminating tumor re-vascularization

Pembrolizumab is a humanized IgG4 kappa monoclonal antibody that blocks the interaction between PD-1 and its ligands, PD-L1 and PD-L2. Pembrolizumab is currently approved for the treatment of unresectable or metastatic melanoma. Analysis of tumor samples before and during treatment in an earlier study demonstrated that a clinical response was associated with an increase in the density of CD8+ T cells in the tumor parenchyma (center), while disease progression was associated with persistent low levels of those cells. In an autochthonous murine model of pancreatic adenocarcinoma, persistent tumor growth despite administration of anti-PD-L1 was similarly associated with failure of tumor-specific cytotoxic T cells to enter the TME despite their presence in the peripheral circulation. This immunosuppressed phenotype was associated with CXCL12 production by cancer-associated fibroblasts. Moreover, administration of a CXCR4 antagonist (AMD3100) induced rapid T-cell accumulation among the cancer cells and, in combination with anti-PD-L1, synergistically decreased tumor growth.

Based on these observations, the hypothesis is that effective CXCR4 antagonism by X4P-001 would be of potential benefit in participants with advanced melanoma and other cancers by multiple mechanisms, resulting in increased anti-tumor immune attack.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a patient must meet all of the following inclusion criteria:

1. Be at least 18 years of age.
2. Has signed the current approved informed consent form.
3. Has a histologically confirmed diagnosis of malignant melanoma.
4. Has at least two separate cutaneous lesions suitable for punch biopsies (at least 3 mm diameter).
5. For women of childbearing potential and men, agree to use a highly effective method of contraceptive from screening, through the study, and for at least 4 weeks after the last dose of study drug.
6. For women of childbearing potential, must have a negative pregnancy test (serum or urine) on Day 1 prior to initiating study treatment, and are not nursing.
7. Be willing and able to comply with the schedule, treatment, and biopsies specified by this protocol.

Exclusion Criteria:

Patients with any of the following will be excluded from participation in the study:

1. Has performance status Grade 2 or higher (Eastern Cooperative Oncology Group [ECOG] criteria).
2. Has ongoing acute clinical adverse events NCI CTCAE Grade 2 or greater resulting from prior cancer therapies (except alopecia).
3. Has had within the past 6 months the occurrence or persistence of one or more of the following medical conditions that could not be controlled with usual medical care (e.g., required emergency care or hospitalization): angina, congestive heart failure, diabetes, seizure disorder.
4. Has had within the past 6 months the occurrence of one or more of the following events: myocardial infarction, cerebrovascular accident, hemorrhage (CTC Grade 3 or 4), chronic liver disease (meeting criteria for Child-Pugh Class B or C), a second active malignancy requiring ongoing treatment during the trial, organ transplantation.
5. Has had within the 4 weeks prior to initiation of study drug, or is expected to have during the study period, surgery requiring general anesthesia
6. Has, at screening, serologic laboratory tests meeting one or more of the following criteria:

   * An indeterminate or positive test for antibody to human immunodeficiency virus (HIV-1 or -2).
   * An indeterminate or positive test for antibody to hepatitis C virus (HCV), unless documented to have no detectable viral load on two independent samples.
   * A positive test for hepatitis B surface antigen (HBsAg).
7. Has, at screening, safety laboratory tests meeting one or more of the following criteria:

   * Hemoglobin <9.0 g/dL
   * Absolute neutrophil count (ANC) <1,500/μL
   * Platelets <100,000/μL
   * Creatinine >2.0x ULN
   * Serum aspartate transaminase (AST) >3x ULN
   * Serum alanine transaminase (ALT) >3x ULN
   * Total bilirubin >1.5x ULN (unless due to Gilbert's Syndrome)
   * International normalized ratio (INR) >1.5x ULN (unless on therapeutic anti-coagulation).
8. Has been previously treated with approved or investigational immunotherapy including oncolytic viruses, or agents directed at CTLA-4, PD-1, or PD-L1 ("checkpoint inhibitors").
9. Has previously received other anti-cancer therapy within 2 weeks prior to Day 1, including radiation therapy or chemotherapy. For investigational anti-cancer therapies, the interval will be determined in consultation with the Medical Monitor.
10. Has, within 2 weeks prior to Day 1, been regularly taking a medication prohibited based on CYP3A4 interaction.
11. Has, at the planned initiation of study drug, an uncontrolled infection.
12. Has any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's successful completion of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Up to 13 weeks, from time of enrollment through study completion or early termination.
Histology Characterization in Sequential Biopsies of Melanoma Lesions | Up to 13 weeks, from time of enrollment through study completion or early termination.

SECONDARY OUTCOMES:
Blood Biomarker Changes | Up to 17 weeks, from time of screening through study completion or early termination.
Minimum Plasma Concentration (Cmin) | Up to 9 weeks, from time of enrollment through end of treatment.
Clinical Tumor Response | Up to 17 weeks, from time of screening through study completion or early termination.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Gan, MD, PhD, Study Director — X4 Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Iowa City, Iowa
  - Clinical Site, Houston, Texas
  - Clinical Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andtbacka RHI, Wang Y, Pierce RH, Campbell JS, Yushak M, Milhem M, Ross M, Niland K, Arbeit RD, Parasuraman S, Bickley K, Yeung CC, Aicher LD, Smythe KS, Gan L. Mavorixafor, an Orally Bioavailable CXCR4 Antagonist, Increases Immune Cell Infiltration and Inflammatory Status of Tumor Microenvironment in Patients with Melanoma. Cancer Res Commun. 2022 Aug 31;2(8):904-913. doi: 10.1158/2767-9764.CRC-22-0090. eCollection 2022 Aug. PMID 36923305